CLINICAL TRIAL: NCT03301285
Title: Study of Efficacy of Zoledronic Acid in the Management of Osteoporosis in Children With Multiple Disabilities
Brief Title: Efficacy of Zoledronic Acid in Osteoporosis of Children With Multiple Disabilities
Acronym: ZOMETA
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: PSS2016/ZOMETA-FEILLET/VS
Record Dates: First submitted 2017-09-21; First posted 2017-10-04 (Actual); Last update posted 2017-10-04 (Actual); Status verified 2017-09

CONDITIONS: Multiple Disability; Osteoporosis
MeSH Terms: conditions — Osteoporosis | interventions — Zoledronic Acid

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children with osteoporosis associated to multiple disabilities: Treated with zoledronic acid
  Interventions: Drug: Zoledronic Acid

INTERVENTIONS:
Drug: Zoledronic Acid — Treatment of osteoporosis

SUMMARY:
The main purpose of this study is the evaluation of the efficacy of zoledronic acid on bone density in children with osteoporosis caused by multiple disabilities.

Secondary purposes are:

1. Description of child population with osteoporosis in the context of motor impairment in Lorraine region
2. Description of osteoporosis stage (level of bone mineralization and clinical consequences) in children with multiple disabilities
3. Description of current osteoporosis preventive care
4. Description of risk factors associated to bone status (drugs)
5. Evaluation of zoledronic acid treatment on fracture numbers
6. Evaluation of zoledronic acid on phosphocalcic profile
7. Description of side effects of zoledronic acid in this indication
8. Description of treatment effects in the sub-population of children with Rett syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Non refusal of parents of participation of their child to the study
* Patients followed for multiple disabilities
* Osteoporosis: lumbar osteodensitometry z-score <-2.5 SD associated or not to pathologic fracture

Exclusion Criteria:

* Bone pathology due to other genetic reasons (rickets, osteogenesis imperfecta)
* Absence of multiple disabilities

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All children followed for osteoporosis associated to multiple disabilities, treated with zoledronic acid, followed at pediatric department of Nancy hospital, between 01/01/2012 and 11/01/2016.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-03-31 (Actual); Study Completion 2017-03-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline (before start of zoledronic acid treatment) lumbar bone density | through study completion, 4 years
  reported in Z-score

SECONDARY OUTCOMES:
Age | Baseline
Sex | Baseline
Height | Baseline
Weight | Baseline
Occurrence of bone fractures | Until baseline
Long-term administration of vitamin/calcium supplement or not | baseline
Administration of drugs or not | baseline
Number of fractures after the start of zoledronic acid treatment | through study completion, 4 years
Change from baseline phosphocalcic profile evaluation | through study completion, 4 years
Frequency of side effects | through study completion, 4 years
Change from baseline lumbar bone density in sub-population of children with Rett syndrome after 1 year of zoledronic acid treatment | 1 year from baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital - CHRU de Nancy, Vandœuvre-lès-Nancy, France

IPD SHARING:
Plan to Share IPD: No